CLINICAL TRIAL: NCT00755105
Title: Body Iron Excretion of Healthy Adults as Measured by Isotope Dilution
Brief Title: Measurements of Body Iron Excretion of Healthy Adults
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC049
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2009-04-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: body iron excretion; Iron isotopes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observation study of subjects who previously had iron-55 isotope administered in studies of iron absorption. By determining the retention of the isotope in blood during a 3-year period, body iron excretion can be measured.

DETAILED DESCRIPTION:
One year following initial administration of iron-55 as a part of other related studies, subjects provide blood samples every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have taken iron-55 in previous study conducted by USDA Grand Forks Human Nutrition Research Center

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult men and women who previously participated in iron absorption studies using iron-55 isotope.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 1998-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet R Hunt, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Derived] Hunt JR, Zito CA, Johnson LK. Body iron excretion by healthy men and women. Am J Clin Nutr. 2009 Jun;89(6):1792-8. doi: 10.3945/ajcn.2009.27439. Epub 2009 Apr 22. PMID 19386738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were invited to join the study if they had participated in a study involving consumption of Iron-55 at least one year earlier at Grand Forks Human Nutrition Research Center
Pre-assignment Details: All enrolled participants were included
Groups:
- Menstruating Women Having Consumed Iron-55 Tracer: Includes women on hormonal contraceptives
Period: Overall Study
Arm/Group | Male Subjects Having Consumed Iron-55 Tracer | Menstruating Women Having Consumed Iron-55 Tracer | Postmenopausal Women Having Consumed Iron-55 Tracer
Started | 38 | 30 | 9
Completed | 29 | 19 | 5
Not Completed | 9 | 11 | 4
Not completed — Withdrawal by Subject | 9 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Male Subjects Having Consumed Iron-55 Tracer | Menstruating Women Having Consumed Iron-55 Tracer | Postmenopausal Women Having Consumed Iron-55 Tracer | Total
Number analyzed (Participants) | 38 | 30 | 9 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (8) | 40 (5) | 50 (5) | 43 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 30 | 9 | 39
  Male | 38 | 0 | 0 | 38

OUTCOME MEASURES:

1. Primary Outcome: Rate of Iron Excretion.
Description: Iron excretion calculated as body Fe (mg) times turnover rate estimated from blood activity of Fe55
Time Frame: 4 years
Population: Per protocol
Measure: Mean (95% Confidence Interval); unit: milligrams per day
Arm/Group | Male Subjects Having Consumed Iron-55 Tracer | Menstruating Women Having Consumed Iron-55 Tracer | Postmenopausal Women Having Consumed Iron-55 Tracer
Number analyzed (Participants) | 29 | 19 | 5
milligrams per day | 1.07 [0.89 to 1.25] | 1.69 [1.30 to 2.20] | 1.08 [0.73 to 1.43]
Statistical Analysis 1: Comparison: Male Subjects Having Consumed Iron-55 Tracer vs Menstruating Women Having Consumed Iron-55 Tracer vs Postmenopausal Women Having Consumed Iron-55 Tracer; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Male Subjects Having Consumed Iron-55 Tracer | Menstruating Women Having Consumed Iron-55 Tracer | Postmenopausal Women Having Consumed Iron-55 Tracer
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/19 | 0/5
Other Adverse Events (participants affected / at risk) | 0/29 | 0/19 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes